CLINICAL TRIAL: NCT06846775
Title: A Case-control Study of the Clinical Utility of DNA Methylation Testing in Patient-collected Vaginal and Urine Samples: A Novel, Patient-friendly and Simple Diagnostic Solution to Detect Endometrial Cancer.
Brief Title: The Clinical Utility of DNA Methylation Testing in Patient-collected Urine and Vaginal Samples to Detect Endometrial Cancer: a Case-control Study
Status: Recruiting | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Central Denmark Region (Other); University of Southern Denmark (Other); Region of Southern Denmark (Other); Amsterdam UMC (Other)
Responsible Party: Sponsor
Other Study IDs: EC-methy-PCS-case-control
Record Dates: First submitted 2025-02-20; First posted 2025-02-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-04

CONDITIONS: Endometrial Cancer
Keywords: DNA-methylation testing; Endometrial Cancer; Patient-collected samples; Urine samples; Vaginal samples
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Patient-collected urine and vaginal samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women with endometrial cancer: Women with diagnosed endometrial cancer ≥ 60 years, without any other concurrent cancer diagnoses. All participants will be asked to collect a urine and vaginal sample, fill out a life style questionnaire and a questionnaire about user experience and preferences.
  Interventions: Diagnostic Test: DNA-methylation testing in patient-collected urine and vaginal samples
- Healthy controls: Gynaecologically and oncolocigally healthy controls ≥ 60 years. All participants will be asked to collect a urine and vaginal sample, fill out a life style questionnaire and a questionnaire about user experience and preferences.
  Interventions: Diagnostic Test: DNA-methylation testing in patient-collected urine and vaginal samples

INTERVENTIONS:
Diagnostic Test: DNA-methylation testing in patient-collected urine and vaginal samples — DNA-methylation testing of methylation markers CDO1, GHSR and ZIC1 for patient-collected vaginal samples and GHSR, CDH13 and SST for patient-collected urine samples.

SUMMARY:
The goal of this observational case-control study is to investigate the use of DNA-methylation testing in patient-collected urine and vaginal samples to detect endometrial cancer. The study aims to answer the following questions:

* Can DNA methylation testing in vaginal and full-void urine samples distinguish endometrial cancer cases from healthy controls?

Researchers will compare patient-collected urine and vaginal samples from patients with diagnosed endometrial cancer (cases) to gynaecologically and oncologically healthy controls (controls).

Participants will

* take a urine and vaginal sample at the hospital.
* answer a questionnaire regarding acceptability and preferences of self-sampling methods.
* answer a lifestyle questionnaire.

DETAILED DESCRIPTION:
BACKGROUND:

Endometrial cancer (EC) incidence is raising and is the fourth most common cancer type in women worldwide with about 417,000 new cases and 90,000 deaths annually. Moreover, EC is the most common gynaecological cancer in developed countries including Denmark with about 800 new cases and 90 deaths yearly. Early diagnosis is essential since the prognosis for women with an advanced EC stage is poor. No screening exists for EC and the most commonly observed clinical symptom is post-menopausal bleeding (PMB), which is a common condition affecting about 11% of postmenopausal women. Because 90% of EC cases are preceded by PMB, referral for specialized gynaecological care through cancer patient pathways is indicated for all Danish women with PMB, causing anxiety among women and high health-care costs. However, only 5-10% of women presenting with PMB have EC.

Worldwide, transvaginal ultrasound (TVUS) evaluation of the endometrium (cut-off: thickness ≥4mm and/or irregular lining of the uterine cavity) is used to identify women with PMB who have the highest cancer risk and therefore require an endometrial biopsy with or without hysteroscopy. While TVUS evaluation is highly sensitive (94.8%) it suffers from low specificity (51%) causing high numbers of unnecessary invasive procedures in healthy women. Moreover, the diagnostic program depends on skilled specialists for ultrasound evaluation, endometrial sampling as well as histopathological examination. This reinforces the clinical urgent and unmet need for a simpler, non-invasive, user-provided and more specific test to aid EC diagnosis.

This study aims to determine whether DNA methylation testing in patient-collected urine and vaginal samples is a clinically safe non-invasive alternative to determine EC risk. Testing for elevated DNA hypermethylation levels of cancer-specific genes has been demonstrated to provide a promising biomarker for detection of early-stage cancers, including cervical and endometrial cancer. DNA hypermethylation has been linked to silencing of tumour suppressor genes, thereby contributing to cancer development. Biologically, the ability to use vaginal and urine material for EC detection by DNA methylation testing is explained by local shedding of EC-derived DNA and cell fragments into the vaginal debris and urine as well as transrenal excretion of tumour-shedded circulating DNA into the urine.

Mainly small proof-of-concepts and case-controls studies have shown feasibility to detect EC using DNA methylation testing in plasma, self-collected vaginal samples, and clinician-collected cervical scrapes. However, the first paper reporting on the diagnostic value of DNA methylation analysis in vaginal samples and urine as a liquid biopsy for EC was just published by co-supervisor Prof. Steenbergen last year. Here, case-control data revealed excellent diagnostic performance of EC-specific DNA methylation markers in patient-collected urine and vaginal samples with sensitivities of 89-90% and specificities of 90-92% for EC detection using markers panels including: CDH13, GHSR, SST, CDO1, and ZIC1.

MATERIALS AND METHODS The vaginal and urine samples will be stored in a biobank at the Dept. of Pathology, Randers Regional Hospital (RHR) until shipment for DNA methylation testing analysis using quantitative methylation-specific PCR (qMSP) in Prof. Steenbergens' laboratory at Amsterdam University Medical Centre, The Netherlands. All samples will be tested for methylation markers, three for vaginal samples (CDO1, GHSR, ZIC1) and three for urine (GHSR, CDH13, SST). Results on endometrial biopsies and hysterectomies including molecular biomarkers and histological type will be retrieved from the nationwide Danish Pathology Databank and the electronic patient journal linked to the patient through the Civil Registration System in Denmark, where all residents have a unique 10-cipher code (CPR-number), to which all health data is linked.

AIM:

1) To determine the diagnostic accuracy of DNA methylation testing in patient-collected full-void urine and vaginal samples to detect EC among cancer cases and healthy controls

RESEARCH PLAN AND FEASIBILITY The study will be conducted in collaboration between University Research Clinic for Cancer Screening, Dept. of Public Health Programmes, Dept. of Pathology, RHR and with gynaecological departments in Central Denmark (Randers and Aarhus) and Southern Denmark Region (Odense) working as inclusion sites. State-of-the-art laboratory facilities are in place at Prof. Steenbergen's laboratory at Amsterdam UMC, supporting the feasibility of the studies.

PERSPECTIVES AND COMMUNICATION If successful, the research will have international impact and result in a novel diagnostic tool that will differentiate between women with PMB who do or do not need specialist referral through cancer patients' pathways to have invasive endometrial biopsies. This will facilitate timely diagnosis, lower the anxiety among patients, and reducing the pressure on the health-care system. Results will be published in international peer-reviewed journals and presented at conferences and will be concluded with a PhD dissertation. The results will be distributed to relevant clinical fora and implemented in national as well as international guidelines.

ELIGIBILITY:
Patients with endometrial cancer (cases): Inclusion Criteria:

* Women ≥ 60 years
* Diagnosed with cancer corpus uteri
* Living in Central Denmark Region or Southern Denmark Region, Denmark
* Able to provide written consent for participation
* Able to read and understand Danish

Patients with endometrial cancer (cases): Exclusion Criteria:

* Other concurrent cancer diagnosis besides cancer corpus uteri
* Withdrawal of consent

Healthy controls: Inclusion Criteria:

* Postmenopausal women ≥ 60 years
* Living in Central Denmark Region, Denmark
* Able to provide written consent for participation
* Able to read and understand Danish

Healthy controls: Exclusion Criteria:

* Diagnosed with cancer or undergoing diagnostic assessment herfore without the last 5 years.
* Vaginal bleeding within the last 3 months.
* Known gynaecological diseases such as cervical dysplasia or atypical endomatrial hyperplasia within the last 5 years.
* Previously hysterectomized
* Withdrawal of consent.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cases will be recruited from Department of Obstetrics and Gynaecology, Aarhus University Hospital, Central Denmark Region, and Odense University Hospital, Southern Denmark Region, Denmark.
  Controls will recruited from Department of Orthopaedics, Randers Regional Hospital, Central Denmark Region, Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
Area Under the Curve | From enrollment and to the end of follow-up at 2 years.
  The diagnostic potential of the six markers for distinguishing patients and controls for EC detection will be illustrated by ROC curves and results will be quantified by AUC with 95% CIs.

CONTACTS AND LOCATIONS:
Overall Officials: Mette Tranberg, Principal Investigator — University Research Clinic for Cancer Screening, Department of Public Health Programmes, Randers Regional Hospital
Locations (3):
- Denmark (3):
  - Department of Obstetrics and Gynaecology, Aarhus University Hospital, Aarhus N
  - Department of Obstetrics and Gynaecology, Odense University Hospital, Odense
  - Department of Orthopaedics, Randers Regional Hospital, Randers

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Erichsen R, Lash TL, Hamilton-Dutoit SJ, Bjerregaard B, Vyberg M, Pedersen L. Existing data sources for clinical epidemiology: the Danish National Pathology Registry and Data Bank. Clin Epidemiol. 2010 Aug 9;2:51-6. doi: 10.2147/clep.s9908. PMID 20865103
- [Background] Evans I, Reisel D, Jones A, Bajrami A, Nijjar S, Solangon SA, Arora R, Redl E, Schreiberhuber L, Ishaq-Parveen I, Rotharmel J, Herzog C, Jurkovic D, Widschwendter M. Performance of the WID-qEC test versus sonography to detect uterine cancers in women with abnormal uterine bleeding (EPI-SURE): a prospective, consecutive observational cohort study in the UK. Lancet Oncol. 2023 Dec;24(12):1375-1386. doi: 10.1016/S1470-2045(23)00466-7. Epub 2023 Nov 6. PMID 37944542
- [Background] Van Keer S, van Splunter AP, Pattyn J, De Smet A, Herzog SA, Van Ostade X, Tjalma WAA, Ieven M, Van Damme P, Steenbergen RDM, Vorsters A. Triage of human papillomavirus infected women by methylation analysis in first-void urine. Sci Rep. 2021 Apr 12;11(1):7862. doi: 10.1038/s41598-021-87329-1. PMID 33846517
- [Background] Guerrero-Preston R, Valle BL, Jedlicka A, Turaga N, Folawiyo O, Pirini F, Lawson F, Vergura A, Noordhuis M, Dziedzic A, Perez G, Renehan M, Guerrero-Diaz C, De Jesus Rodriguez E, Diaz-Montes T, Rodriguez Orengo J, Mendez K, Romaguera J, Trock BJ, Florea L, Sidransky D. Molecular Triage of Premalignant Lesions in Liquid-Based Cervical Cytology and Circulating Cell-Free DNA from Urine, Using a Panel of Methylated Human Papilloma Virus and Host Genes. Cancer Prev Res (Phila). 2016 Dec;9(12):915-924. doi: 10.1158/1940-6207.CAPR-16-0138. Epub 2016 Sep 26. PMID 27671338
- [Background] Snoek BC, Splunter APV, Bleeker MCG, Ruiten MCV, Heideman DAM, Rurup WF, Verlaat W, Schotman H, Gent MV, Trommel NEV, Steenbergen RDM. Cervical cancer detection by DNA methylation analysis in urine. Sci Rep. 2019 Feb 28;9(1):3088. doi: 10.1038/s41598-019-39275-2. PMID 30816167
- [Background] Wever BMM, van den Helder R, van Splunter AP, van Gent MDJM, Kasius JC, Trum JW, Verhoeve HR, van Baal WM, Hulbert A, Verhoef L, Heideman DAM, Lissenberg-Witte BI, van Trommel NE, Steenbergen RDM, Bleeker MCG. DNA methylation testing for endometrial cancer detection in urine, cervicovaginal self-samples and cervical scrapes. Int J Cancer. 2023 Jul 15;153(2):341-351. doi: 10.1002/ijc.34504. Epub 2023 Mar 23. PMID 36912267
- [Background] Bakkum-Gamez JN, Sherman ME, Slettedahl SW, Mahoney DW, Lemens MA, Laughlin-Tommaso SK, Hopkins MR, VanOosten A, Shridhar V, Staub JK, Cao X, Foote PH, Clarke MA, Burger KN, Berger CK, O'Connell MC, Doering KA, Podratz KC, DeStephano CC, Schoolmeester JK, Kerr SE, Wentzensen N, Taylor WR, Kisiel JB. Detection of endometrial cancer using tampon-based collection and methylated DNA markers. Gynecol Oncol. 2023 Jul;174:11-20. doi: 10.1016/j.ygyno.2023.04.014. Epub 2023 May 2. PMID 37141817
- [Background] De Strooper LM, van Zummeren M, Steenbergen RD, Bleeker MC, Hesselink AT, Wisman GB, Snijders PJ, Heideman DA, Meijer CJ. CADM1, MAL and miR124-2 methylation analysis in cervical scrapes to detect cervical and endometrial cancer. J Clin Pathol. 2014 Dec;67(12):1067-71. doi: 10.1136/jclinpath-2014-202616. Epub 2014 Oct 3. PMID 25281766
- [Background] Kim GE, Kweon SS, Lee JS, Lee JH, Nam JH, Choi C. Quantitative assessment of DNA methylation for the detection of cervical and endometrial adenocarcinomas in liquid-based cytology specimens. Anal Quant Cytopathol Histpathol. 2012 Aug;34(4):195-203. PMID 23016466
- [Background] Doufekas K, Hadwin R, Kandimalla R, Jones A, Mould T, Crowe S, Olaitan A, Macdonald N, Fiegl H, Wik E, Salvesen HB, Widschwendter M. GALR1 methylation in vaginal swabs is highly accurate in identifying women with endometrial cancer. Int J Gynecol Cancer. 2013 Jul;23(6):1050-5. doi: 10.1097/IGC.0b013e3182959103. PMID 23727823
- [Background] Fiegl H, Gattringer C, Widschwendter A, Schneitter A, Ramoni A, Sarlay D, Gaugg I, Goebel G, Muller HM, Mueller-Holzner E, Marth C, Widschwendter M. Methylated DNA collected by tampons--a new tool to detect endometrial cancer. Cancer Epidemiol Biomarkers Prev. 2004 May;13(5):882-8. PMID 15159323
- [Background] den Helder RV, Wever BM, van Trommel JA, Ket JC, Bleeker MC, Steenbergen RD, van Trommel NE. DNA methylation markers for endometrial cancer detection in minimally invasive samples: a systematic review. Epigenomics. 2020 Sep;12(18):1661-1672. doi: 10.2217/epi-2020-0164. Epub 2020 Sep 17. PMID 32938224
- [Background] Hentschel AE, van den Helder R, van Trommel NE, van Splunter AP, van Boerdonk RAA, van Gent MDJM, Nieuwenhuijzen JA, Steenbergen RDM. The Origin of Tumor DNA in Urine of Urogenital Cancer Patients: Local Shedding and Transrenal Excretion. Cancers (Basel). 2021 Jan 31;13(3):535. doi: 10.3390/cancers13030535. PMID 33572525
- [Background] Kulis M, Esteller M. DNA methylation and cancer. Adv Genet. 2010;70:27-56. doi: 10.1016/B978-0-12-380866-0.60002-2. PMID 20920744
- [Background] van den Helder R, Wever BMM, van Trommel NE, van Splunter AP, Mom CH, Kasius JC, Bleeker MCG, Steenbergen RDM. Non-invasive detection of endometrial cancer by DNA methylation analysis in urine. Clin Epigenetics. 2020 Nov 3;12(1):165. doi: 10.1186/s13148-020-00958-7. PMID 33143739
- [Background] Morice P, Leary A, Creutzberg C, Abu-Rustum N, Darai E. Endometrial cancer. Lancet. 2016 Mar 12;387(10023):1094-1108. doi: 10.1016/S0140-6736(15)00130-0. Epub 2015 Sep 6. PMID 26354523
- [Background] Herzog C, Marin F, Jones A, Evans I, Reisel D, Redl E, Schreiberhuber L, Paytubi S, Pelegrina B, Carmona A, Peremiquel-Trillas P, Frias-Gomez J, Pineda M, Brunet J, Ponce J, Matias-Guiu X, de Sanjose S, Alemany L, Olaitan A, Wong M, Jurkovic D, Crosbie EJ, Rosenthal AN, Bjorge L, Zikan M, Dostalek L, Cibula D, Sundstrom K, Dillner J, Costas L, Widschwendter M. A Simple Cervicovaginal Epigenetic Test for Screening and Rapid Triage of Women With Suspected Endometrial Cancer: Validation in Several Cohort and Case/Control Sets. J Clin Oncol. 2022 Nov 20;40(33):3828-3838. doi: 10.1200/JCO.22.00266. Epub 2022 Aug 24. PMID 36001862
- [Background] Astrup K, Olivarius Nde F. Frequency of spontaneously occurring postmenopausal bleeding in the general population. Acta Obstet Gynecol Scand. 2004 Feb;83(2):203-7. doi: 10.1111/j.0001-6349.2004.00400.x. PMID 14756741
- [Background] Long B, Clarke MA, Morillo ADM, Wentzensen N, Bakkum-Gamez JN. Ultrasound detection of endometrial cancer in women with postmenopausal bleeding: Systematic review and meta-analysis. Gynecol Oncol. 2020 Jun;157(3):624-633. doi: 10.1016/j.ygyno.2020.01.032. Epub 2020 Jan 31. PMID 32008795
- [Background] Gustafson LW, Booth BB, Kahlert J, Ortoft G, Mejlgaard E, Clarke MA, Wentzensen N, Rositch AF, Hammer A. Trends in hysterectomy-corrected uterine cancer mortality rates during 2002 to 2015: mortality of nonendometrioid cancer on the rise? Int J Cancer. 2021 Feb 1;148(3):584-592. doi: 10.1002/ijc.33219. Epub 2020 Aug 17. PMID 32683690
- [Background] Engholm G, Ferlay J, Christensen N, Bray F, Gjerstorff ML, Klint A, Kotlum JE, Olafsdottir E, Pukkala E, Storm HH. NORDCAN--a Nordic tool for cancer information, planning, quality control and research. Acta Oncol. 2010 Jun;49(5):725-36. doi: 10.3109/02841861003782017. PMID 20491528
- [Background] Lu KH, Broaddus RR. Endometrial Cancer. N Engl J Med. 2020 Nov 19;383(21):2053-2064. doi: 10.1056/NEJMra1514010. No abstract available. PMID 33207095
- [Background] Crosbie EJ, Kitson SJ, McAlpine JN, Mukhopadhyay A, Powell ME, Singh N. Endometrial cancer. Lancet. 2022 Apr 9;399(10333):1412-1428. doi: 10.1016/S0140-6736(22)00323-3. PMID 35397864
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338